CLINICAL TRIAL: NCT05991752
Title: Evaluation médico-économique du Diagnostic précoce Des récidives de Cancer épithélial Ovarien Par le Score ROMA : Essai Prospectif Multicentrique randomisé
Brief Title: Health-Economic Evaluation of Early Diagnosis of Epithalial Ovarian Cancer Recurrence Using the ROMA Score: a Prospective Multicenter Randomized Trial
Acronym: ROMECO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DR210313
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROMA Score (Experimental): Experimental group: CA125 and HE4 assays every 4 months for 3 years to assess the ROMA score, in addition to the recommended conventional follow-up.
  Interventions: Diagnostic Test: ROMA score evaluation
- CA125 alone (No Intervention): Control group: CA125 assay alone every 4 months for 3 years, as part of the recommended standard follow-up.

INTERVENTIONS:
Diagnostic Test: ROMA score evaluation — Every 4 months, for 3 years, patients in the experimental group will done a biological examination based on assessment of the ROMA score (CA125+HE4 assay).
  Arms: ROMA Score

SUMMARY:
In this study, we hypothesize that calculating the ROMA score (CA125 + HE4 blood marker assay) will enable faster, more targeted diagnosis and management of epithelial ovarian cancer recurrence than the CA125 marker assay alone. This early identification of recurrence would then improve patients' quality of life, since it would increase the chances of benefiting from less invasive and less morbid surgery. It would also reduce the cost of patient management following disease progression. If our hypothesis is confirmed, the results of this study will enable us to update the recommendations for post-treatment follow-up of patients in remission from epithelial ovarian cancer, as well as reimbursing the HE4 marker assay (and thus the calculation of the ROMA score).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or over and less than 85 years old
* With proven FIGO stage I to IV epithelial ovarian cancer (ovary/tumor/peritoneum)
* Women in remission after first-line chemotherapy, with a normal CA125 less than 4 months old at study entry (end of first-line chemotherapy).
* Woman having completed chemotherapy at least 6 months previously
* Written informed consent
* French social security

Exclusion Criteria:

* Any physical or psychiatric condition that may interfere with the patient's cooperation in data collection
* Patient with normal CA125 at initial diagnosis of epithelial ovarian cancer
* Patient under guardianship
* Patient deprived of liberty

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 320 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Incremental Cost-Utility Ratio (ICUR) expressed as the cost per QALY gained at 36 months of using the ROMA score compared to usual follow-up with the CA-125 test, from the collective perspective. | 36 months
  QALYs (Quality-Adjusted Life Years) will be estimated from patient responses to the EQ-5D-5L instrument (EuroQol group - 5 Dimensions - 5 levels). The cost evaluation will identify, measure and value all the resources consumed in the production of overall care: hospital and outpatient care, transport, informal care, and social aid services. All consumed resources will be estimated from the collective perspective. QALY and cost data will be used to estimate this within-trial ICUR.

SECONDARY OUTCOMES:
Incremental Cost-Effectiveness Ratio (ICER) expressed as the cost per life-year gained at 36 months of using the ROMA score compared to usual follow-up with the CA-125 test, from the collective perspective. | 36 months
  Cost and survival data will be used to estimate the within-trial ICER.
Incremental Cost-Utility Ratio (ICUR) expressed as the cost per QAPFY gained at 36 months of using the ROMA score compared to usual follow-up with the CA-125 test, from the collective perspective. | 36 months
  QAPFY (Quality-Adjusted Progression-Free Years) will be estimated using the progression-free survival data and patient responses to the EQ-5D-5L instrument. Cost and QAPFY data will be used to estimate this within-trial ICUR.
Financial impact per year and over a 5-year period of spreading the use of the ROMA score in the routine follow-up of patients for the diagnosis of the first recurrence of epithelial ovarian cancer. | per year and over a 5-year period
  The financial impact will be estimated from the French Health Insurance, using a budget impact model.
Characteristics of recurrence between the two groups (i.e. time to recurrence, location and operability) | 36 months
  Proportion of patients with a first operable recurrence, median interval between randomization and diagnosis of recurrence by imaging or biopsy
Characteristics of treatments for first recurrence (including surgery) | 36 months
  Proportion of patients with complete surgery without macroscopic residue, without reoperation, proportion of other therapies: chemotherapy/hormone therapy/other therapies
Quality of life of women | 36 months
  Quality of life assessed by the EORTC QLQ-C30 and EORTC QLQ-OV28 (European Organization for Research and Treatment in Cancer Quality Life Questionnaire) every 4 months for 3 years
Evolution of CA125, HE4 and ROMA score after management of the first recurrence | 36 months
  Description of the evolution of CA125, HE4 and ROMA score after management of the first recurrence
Estimation and validation of a mapping function from the specific EORTC QLQ-C30 and EORTC QLQ-OV28 questionnaires to the generic EQ-5D5L questionnaire. | 36 months
  Deriving the EQ5D-5L score from responses to the EORTC QLQ-C30 and QLQ-OV28 questionnaires in women undergoing post-treatment remission follow-up of epithelial ovarian cancer.